CLINICAL TRIAL: NCT04497727
Title: Gut Inflammation and Gut-Gut Microbiome Interactions in the Pathogenesis of Hypertension
Brief Title: Gut Organoid and Microbiome Interactions in Hypertension
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201903360 -N; R01HL132448 (NIH)
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Results first posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Gut Inflammation; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Gene Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During your scheduled colonoscopy, a maximum of 4 biopsies will be taken from your colon.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing routine colonoscopy: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent. Based on their blood pressure status, participants were categorized into two groups: individuals without hypertension (normotensive group) and individuals with high blood pressure (hypertensive group), defined according to the 2017 ACC/AHA guidelines
  Interventions: Other: Gene Expression

INTERVENTIONS:
Other: Gene Expression — Gene expression analysis of biopsy specimens obtained during routine colonoscopy examination

SUMMARY:
The study compared basic properties of gut epithelia of hypertensive and normotensive reference subjects. The study determined if there are fundamental differences in the gut epithelium in hypertension compared to normotension. Specifically, this study examined gene expression profiles of gut organoids derived from biopsy samples of hypertensive and normotensive individuals undergoing clinically indicated colonoscopy.

DETAILED DESCRIPTION:
This investigated whether there is a difference in gut epithelia between individuals with and without high blood pressure by comparing colonic biopsy samples from. The study was conducted among adults undergoing routine elective colonoscopy at the University of Florida. Participants were classified into high blood pressure (HBP) and normotensive (REF) groups based on blood pressure criteria defined by the 2017 ACC/AHA guidelines.

The study had two primary aims. Aim 1 was to evaluate whether gene expression patterns in the gut epithelium differ between hypertensive and normotensive individuals using RNA sequencing. Aim 2 was to assess whether gut organoids-three-dimensional epithelial cultures derived from colonic biopsies-exhibit different growth rates and proportions, using immunohistochemistry and fluorescence-activated cell sorting (FACS).

Biopsy specimens were collected during clinically indicated colonoscopies. Tissue samples were processed immediately after collection: one portion was snap-frozen for RNA isolation and sequencing; the other was used to establish gut organoid cultures. Data were coded and stored in a secure, encrypted database with all identifiers removed to protect confidentiality, in compliance with HIPAA regulations.

Although the study protocol initially planned to recruit 60 participants, a total of 35 subjects were successfully enrolled-16 with high blood pressure (HBP) and 19 normotensive (REF) participants. All provided adequate biopsy material for gene expression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion/exclusion criteria for hypertension participants
* Ages: 18-80 years old with a weight greater than or equal to 110 lbs
* Diagnosis of hypertension or without hypertension for the reference cohort. 2017 ACC/AHA (American College of Cardiology/American Heart Association) definition for hypertension (systolic blood pressure ≥130 mmHg and/or diastolic BP ≥80 mmHg) will be used.
* Scheduled elective colonoscopy

Exclusion Criteria:

* Hypertensive or reference individuals with history of autoimmune disease or other chronic inflammatory conditions.
* Pregnant or have been pregnant in the last six months.
* Antibiotic treatment within two months of study enrollment
* Currently taking a medication (e.g. antibiotic, anti-inflammatory agents, glucocorticoids, other immune modulating medications, antacids or proton pump inhibitor drugs like Prilosec) known to modify gut microbiota.
* Unwilling to discontinue using probiotics for at least two weeks before scheduled biopsy.
* History of intestinal surgery, inflammatory bowel disease, celiac disease, lactose intolerance, chronic pancreatitis or other malabsorption disorder.
* History of blood transfusion within 4 weeks.
* Subjects who, in the opinion of the investigator, will be uncooperative or unable to comply with study procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hypertensive and normotensive patients who routinely undergo scheduled elective colonoscopy (for different, not selected reasons)
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2024-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Pepine, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertensive Group: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent. Based on their blood pressure status, participants were categorized as individuals with high blood pressure (hypertensive group), defined according to the 2017 ACC/AHA guidelines
- Normotensive Group: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent. Based on their blood pressure status, participants were categorized as individuals without hypertension (normotensive group) defined according to the 2017 ACC/AHA guidelines
  Gene Expression: Gene expression analysis of biopsy specimens obtained during routine colonoscopy examination
Period: Overall Study
Arm/Group | Hypertensive Group | Normotensive Group
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypertensive Group: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent. Based on their blood pressure status, participants were categorized as individuals with high blood pressure (hypertensive group), defined according to the 2017 ACC/AHA guidelines
  Gene Expression: Gene expression analysis of biopsy specimens obtained during routine colonoscopy examination
- Normotensive Group: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent. Based on their blood pressure status, participants were categorized as individuals without hypertension (normotensive group), defined according to the 2017 ACC/AHA guidelines
- Total: Total of all reporting groups
Arm/Group | Hypertensive Group | Normotensive Group | Total
Number analyzed (Participants) | 16 | 19 | 35
Age, Continuous [Mean (Inter-Quartile Range); unit: Years] | 62 [57 to 68] | 55 [50 to 60] | 58 [53 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: Participants]
  United States | 16 | 19 | 35

OUTCOME MEASURES:

1. Primary Outcome: Differential Gene Expression in Gut Epithelium
Description: Number of differentially expressed genes identified through RNA sequencing of colonic epithelial tissue obtained during colonoscopy. Expression profiles were compared between individuals with High Blood pressure (HBP) (hypertensive group) and normotensive reference (REF) participants. Genes were considered differentially expressed if they met criteria of false discovery rate (FDR)-adjusted p-value < 0.05 and absolute fold change ≥ 1.5.
Time Frame: At time of colonoscopy (single visit)
Population: Colonic biopsies from HBP participants revealed 35 differentially expressed genes (29 upregulated, 6 downregulated) compared to normotensive subjects (reference group).
Measure: Number; unit: Differentially expressed gene
Groups:
- All Study Participants: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent.
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
Differentially expressed gene
  Upregulated Genes | 29
  Downregulated Genes | 6

2. Primary Outcome: Growth Rates of Gut Organoids
Description: To compare growth rates and proportions of gut organoids derived from High Blood pressure (HBP) vs. normotensive (REF) participants.
Time Frame: Within days to weeks post-biopsy (in vitro culture period)
Population: No data obtained for this outcome measure because organoid preparations did not meet feasibility criteria for sample quantity and quality required for FACS and IHC. Further samples will never be obtained.
Arm/Group | Patients Undergoing Routine Colonoscopy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From time of colonoscopy procedure through discharge from the recovery area, for an average total duration of approximately 60 minutes.
Groups:
- Normotensive Group: Participants were adults undergoing routine screening colonoscopy who met study eligibility criteria and provided written informed consent. Based on their blood pressure status, participants were categorized as individuals without hypertension (normotensive group), defined according to the 2017 ACC/AHA guidelines
  Gene Expression: Gene expression analysis of biopsy specimens obtained during routine colonoscopy examination
Arm/Group | Hypertensive Group | Normotensive Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/19
Other Adverse Events (participants affected / at risk) | 0/16 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/27/NCT04497727/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT04497727/ICF_000.pdf